CLINICAL TRIAL: NCT07087795
Title: A Study to Investigate Efficacy and Safety of NNC0194-0499 Versus Placebo, Both Administered Alone or in Combination With Semaglutide in People With Type 1 Diabetes
Brief Title: A Study to See the Effect of NNC0194-0499 Alone or in Combination With Semaglutide on Blood Sugar Control in People Living With Type 1 Diabetes
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN6497-8316; U1111-1315-5122 (Other: World Health Organization (WHO)); 2024-519533-38 (Other: European Medical Agency (EMA))
Record Dates: First submitted 2025-06-29; First posted 2025-07-28 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part A: NNC0194-0499/Placebo (Experimental): After a 2-week run-in period; participants will be randomised 1:1 to a treatment sequence with two 7-week treatment periods of once weekly subcutaneous NNC0194-0499 or placebo. Between the two treatment periods; there is a wash-out period. After the wash-out period, there will be a cross over, ensuring that all the participants receive both NNC0194-0499 and placebo.
  Interventions: Drug: NNC0194-0499; Drug: Placebo
- Part B: NNC0194-0499/Placebo + Semaglutide (Experimental): After the 2-week run-in phase followed by the 8-week of dose escalation period (every 4 weeks) of once weekly subcutaneous semaglutide; participants will be randomised 1:1 to a treatment sequence with two 7-week treatment periods of once weekly subcutaneous NNC0194-0499 or placebo and continued semaglutide. Between the two treatment periods; there is a wash-out period where the participant continues to receive once weekly subcutaneous semaglutide. After the wash-out period, there will be a cross over, ensuring that all the participants receive both NNC0194-0499 and placebo together with semaglutide.
  Interventions: Drug: NNC0194-0499; Drug: Placebo; Drug: Semaglutide

INTERVENTIONS:
Drug: NNC0194-0499 — Participants will receive subcutaneous NNC0194-0499 once weekly.
Drug: Placebo — Participants will receive placebo matched to NNC0194-0499 subcutaneously.
Drug: Semaglutide — Participants will receive subcutaneous semaglutide once weekly.
  Arms: Part B: NNC0194-0499/Placebo + Semaglutide

SUMMARY:
This study is testing the effect of a new study medicine NNC0194-0499 in type 1 diabetes. The purpose of the study is to compare the effect of NNC0194-0499 on the blood sugar levels of participants with type 1 diabetes when taken in combination with semaglutide or placebo. All participants will receive standard of care insulin treatment. The study will last for about 36 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male or female.
* Age 18-64 years (both inclusive) at the time of signing the informed consent.
* Body mass index 22-35 kilogram per square meter (kg/m^2) (both inclusive) for Part A and 27-35(kg/m^2) (both inclusive) for Part B at the day of screening.
* Diagnosed with type 1 diabetes mellitus greater than equal to (≥) 1 year prior to the day of screening.
* Treated with multiple daily insulin injections and stable insulin dose greater than (>) 90 days prior to the day of screening, as judged by the investigator.
* Use of Continuous glucose monitoring (CGM) device > 180 consecutive days prior to the day of screening.
* Glycated haemoglobin (HbA1c) from 7.2 - 9.0% (both inclusive).
* Considered to be generally healthy (except for mild conditions under stable treatment associated with type 1 diabetes mellitus) based on the medical history, physical examination, and the results of vital signs, electrocardiogram and clinical laboratory tests performed during the screening visit, as judged by the investigator.
* Ability and willingness to wear the Novo Nordisk provided CGM device according to the protocol including replacement of CGM sensor at home.
* Ability and willingness to refrain from wearing own CGM/Flash glucose monitor for the duration of the study, as judged by the investigator.

Exclusion Criteria:

* Any condition, except for mild conditions under stable treatment associated with type 1 diabetes mellitus, which in the investigator's opinion might jeopardise participant's safety or compliance with the protocol.
* Treatment with glucagon-like peptide-1(GLP-1) RA within 90 days before screening.
* Use of any medication with unknown or unspecified content within 90 days before screening.
* Presence or history of cardiovascular disease including stable and unstable angina pectoris, myocardial infarction, transient ischaemic attack, stroke, cardiac decompensation, clinically significant arrhythmias or clinically significant conduction disorders.
* Presence or history of any clinically relevant respiratory, metabolic, renal, hepatic, gastrointestinal, endocrinological conditions (except conditions associated with diabetes mellitus and obesity).
* Recurrent severe hypoglycaemia (more than 1 severe hypoglycaemic event within 180 days) or hypoglycaemic unawareness as judged by the investigator or hospitalisation for diabetic ketoacidosis within 180 days prior to the day of screening.
* Any episode of diabetic ketoacidosis within 90 days before screening.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 96 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-09-12 (Estimated); Study Completion 2026-09-25 (Estimated)

PRIMARY OUTCOMES:
Part A: Change in time in range (TIR) 3.9-10.0 mmol/L (70-80 mg/dL) | From baseline (day -14 - -1) to day 36-49 / day 106-119
  Percentage point (%-points).
Part B: Change in time in range (TIR) 3.9-10.0 mmol/L (70-80 mg/dL) | From baseline (day -14 - -1) to day 92-105 / day 162-175
  %-points.

SECONDARY OUTCOMES:
Change in coefficient of variation (CV) of sensor glucose, total | Part A: From baseline (day -14 - -1) to day 36-49 / day 106-119; Part B: From baseline (day -14 - -1) to day 92-105 / day 162-175
  %-points.
Change in mean sensor glucose (SG) | Part A: From baseline (day -14 - -1) to day 36-49 / day 106-119; Part B: From baseline (day -14 - -1) to day 92-105 / day 162-175
  Millimoles per liter (mmol/L).
Change in time above range (TAR) >10.0 mmol/L (>180 mg/dL) | Part A: From baseline (day -14 - -1) to day 36-49 / day 106-119; Part B: From baseline (day -14 - -1) to day 92-105 / day 162-175
  %-points.
Change in time above range (TAR) >13.9 mmol/L (>250 mg/dL) | Part A: From baseline (day -14 - -1) to day 36-49 / day 106-119; Part B: From baseline (day -14 - -1) to day 92-105 / day 162-175
  %-points.
Time below range (TBR) <3.9 mmol/L (70 mg/dL) | Part A: day 36-49/ day 106-119; Part B: day 92-105/ day 162-175
  % of time.
Time below range (TBR)<3.0 mmol/L (54 mg/dL) | Part A: day 36-49/ day 106-119; Part B: day 92-105/ day 162-175
  % of time.
Change in time in tight range (TITR) 3.9-7.8 mmol/L (70-140 mg/dL) | Part A: From baseline (day -14 - -1) to day 36-49 / day 106-119; Part B: From baseline (day -14 - -1) to day 92-105 / day 162-175
  %-points.
Change in mean total daily insulin dose per kg | Part A: From baseline (day -3 - -1) to day 36-49 / day 106-119; Part B: From baseline (day -3 - -1) to day 92-105 / day 162-175
  Ratio to baseline.
Change in triglycerides | Part A: From baseline (day 1) to day 50/ day 120; Part B: From baseline (day 1) to day 106/ day 176
  Ratio to baseline.
Number of adverse events (AEs) | Part A: From baseline (day 1) to day 155; Part B: From baseline (day 1) to day 211
  Number of events.
Number of severe hypoglycaemic episodes (level 3) | Part A: From baseline (day 1) to day 155; Part B: From baseline (day 1) to day 211
  Number of episodes.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (1):
- Profil Institut für Stoffwechselforschung GmbH, Neuss, Germany

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com.
URL: http://novonordisk-trials.com